CLINICAL TRIAL: NCT04049903
Title: A First-In-Human, Single-Arm, Multi-Center, Open-Label, Repeated-Dose, Dose-Escalation Study of MP0310 in Patients With Advanced Solid Tumors
Brief Title: Study to Investigate the Safety, Blood Levels and Activity of MP0310 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Molecular Partners AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MP0310-CP101; 2018-004786-13 (EudraCT Number)
Record Dates: First submitted 2019-08-05; First posted 2019-08-08 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MP0310 Part A (Experimental): Enrollment will follow a standard 3 + 3 dose escalation design. Sequential Cohorts of patients will be dosed until the MTD or unacceptable toxicity is reached. Up to 12 additional patients in total may be included at selected dose levels (up to 3).
  Interventions: Drug: MP0310
- MP0310 Part B (Experimental): weekly schedule, at least 3 and up to 24 patients evaluable for DLT assessment will be enrolled (1 to 4 cohorts with 3 to 6 patients each (3 initial plus up to 3 backfill patients)).
  Interventions: Drug: MP0310
- MP0310 Part C (Experimental): q3w schedule implementing B-cell depletion, at least 3 and up to 12 patients evaluable for DLT assessment will be enrolled (1 to 2 cohorts with 3 to 6 patients each (3 initial plus up to 3 backfill patients)).
  Interventions: Drug: MP0310

INTERVENTIONS:
Drug: MP0310 — MP0310 will be examined for safety, tolerability, PK, and PD activity in subjects with advanced solid tumors

SUMMARY:
To evaluate the safety and tolerability of MP0310, a DARPin® therapeutic candidate for tumor targeted activation of T cells, in patients with advanced solid tumors

ELIGIBILITY:
Inclusion criteria:

1. Patient has an advanced, histologically-proven solid tumor of one of the following types, treated with at least one line of systemic therapy, and for which approved therapies have been exhausted or for which the Investigator considers the patient ineligible or intolerant of other forms of treatment: Colorectal, Ovarian, Endometrial, Gastric, Pancreatic, Anal, Cervical, Squamous cell cancer of the head and neck, Mesothelioma, Prostate, Non-small cell lung cancer, Melanoma, Urothelial/bladder, Microsatellite instability high tumors of any type, Cutaneous squamous cell, Breast,
2. Patients have to be willing to comply with study procedures
3. ≥18 years of age
4. Mentally competent, able to understand and willing to sign the ICF
5. Eastern Cooperative Oncology Group performance status (ECOG; PS) ≤1
6. Anticipated life expectancy ≥12 weeks by Investigator judgment
7. The disease is measurable according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria
8. Mandatory paired pre- and on-treatment biopsies - preferably from the same lesion - are required as follows:

   1. At least 1 tumor lesion ≥10 mm amenable to percutaneous biopsy other than the target lesion used to follow response as defined by RECIST v1.1
   2. For cutaneous or subcutaneous lesions, tumors should be ≥ 5mm in diameter amenable to paired biopsy by excisional or punch biopsies without unacceptable risk of a major procedural complication
   3. For core needle biopsy specimens three to six 18 gauge cores should be collected. If more than 1 biopsy is planned to be taken from one lesion, the lesion should be large enough to permit successive biopsies preferably ≥1 cm apart.
9. At least 4 weeks must have elapsed from any prior major surgery. The following procedures are not considered major surgical procedure:

   1. Obtaining the pre-treatment biopsy as per protocol requirements
   2. Placement of a port for central venous access
   3. Needle, punch or excisional biopsy of a clinically or radiographically detected lesion
10. Laboratory values at screening must be:

    a. Adequate hematology: i. platelet count ≥100,000 cells/mm3 ii. absolute neutrophil count ≥1,000 cells/mm3 iii. hemoglobin ≥9 g/dL b. Serum creatinine ≤1.5 x upper limit of normal (ULN) or creatinine clearance ≥50 mL/min on the basis of CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration), Cockcroft-Gault, or Modification of Diet in Renal Disease (MDRD) glomerular filtration rate estimation c. Adequate coagulation: iv. INR must be <1.5, unless on therapeutic anticoagulants v. PT and activated partial thromboplastin time (aPTT) ≤1.6 x ULN unless therapeutically warranted d. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <3x ULN e. Bilirubin <1.5 x ULN, except for patients with a known familial hyperbilirubinemia (such as e.g., Gilbert syndrome). For patients with documented Gilbert's syndrome (Gilbert-Meulengracht syndrome) total bilirubin <3 x ULN is acceptable) f. Potassium, calcium, and magnesium that are >0.9 of LLN and ≤1.1 of ULN. Supplementation is allowed for potassium, calcium and magnesium to reach these values
11. A woman of childbearing potential (WOCBP) should only be included after a confirmed menstrual period and a negative serum pregnancy test at Screening.

    a. Where ovarian activity is being suppressed by chemotherapy, confirmation of non-pregnancy by menstrual period is not required
12. A female patient is eligible to participate if she is not pregnant, not breastfeeding (for 12 months following last dose of rituximab), and at least one of the following conditions applies:

    1. Not a woman of child bearing potential (WOCBP)
    2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 3 months after the last dose of MP0310 and 12 months after the last dose of rituximab, whichever is longer.
13. Men who are not surgically sterilized (and with appropriate post vasectomy documentation of the absence of sperm in the ejaculate) and who are partners of WOCBP must be willing to use adequate contraception as detailed in Section 15.7 from the Screening visit, during the treatment period, and for at least 3 months after the last MP0310 IMP administration and refrain from donating sperm during this period.
14. Covered by healthcare insurance (if applicable, in accordance with local regulations)

Exclusion criteria

1. Known hypersensitivity to the following excipients that are used for formulation of MP0310:

   a. L-histidine, L-histidine hydrochloride, D-mannitol and polysorbate 20
2. Patients with autoimmune diseases, except auto-immune endocrinopathies that are stable with hormone replacement therapy
3. Patients with inflammatory diseases such as arthritis, colitis, liver fibrosis, cirrhosis, interstitial fibrosis, or COPD (chronic obstructive pulmonary disease; that may have elevated tissue FAP expression) unless approved after consultation by the Medical Monitor (MM).
4. Concurrent enrollment in another clinical study, unless it is an observational (non interventional) clinical study for the duration of this study or the follow-up period of an interventional study
5. Patient was previously treated in this study
6. Serious illness or concomitant non-oncological disease considered by the Investigator to be incompatible with participating in the protocol
7. Bisphosphonate therapy for symptomatic hypercalcemia

   a. Patients on stable dose of bisphosphonate therapy or receptor activator of nuclear kappa-B ligand (RANKL)-therapy for more than 8 weeks prior to first scheduled dose of MP0310 for other reasons (e.g., bone metastasis or osteoporosis) are allowed
8. Use of an investigational agent within the past 4 weeks before first MP0310 IMP administration in this study
9. Any anti-cancer therapy, including chemotherapy, hormonal therapy, or radiotherapy, within 3 weeks prior to first MP0310 IMP administration; however, the following are allowed:

   1. Hormonal therapy with gonadotropin-releasing hormone (GnRH) agonists or antagonists for prostate cancer
   2. Hormone-replacement therapy or oral contraceptives
   3. Palliative radiotherapy for bone metastases 2 weeks prior to first MP0310 IMP administration
10. Corticosteroid use exceeding 10 mg/day prednisone or equivalent
11. Left ventricular ejection fraction of <50% on echocardiographic exam or multigated acquisition (MUGA) scan at screening
12. Any history or evidence of clinically significant cardiovascular disease defined as at least one of the following criteria:

    1. Evidence of poorly controlled arterial hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg)
    2. Myocardial infarction or instable angina pectoris within the previous 6 months
    3. Documented history of congestive heart failure of New York Heart Association >2 criteria
    4. Any cardiac arrhythmia that is not well controlled
    5. QT corrected (QTc) prolongation > Grade 1 (>480 ms) at screening measured on 2 separate electrocardiograms (ECGs) at least 10 minutes apart
    6. Clinically significant valvular heart disease
13. Severe dyspnea, pulmonary dysfunction, or need for continuous supportive oxygen inhalation
14. Arterial thromboembolic event, stroke, or transient ischemia attack within the past 12 months
15. Patients with known central nervous system (CNS) metastasis that are either untreated or are treated but are associated with clinical symptoms (e.g., headache, convulsions). Patients with CNS metastasis that have been treated with radiotherapy and/or surgery are eligible if they are clinically without symptoms for at least 6 weeks; if under treatment with corticosteroids (not exceeding 10 mg/day prednisone or equivalent) and/or anticonvulsive agents patients must be on a stable dose for at least two weeks.
16. Any active uncontrolled bleeding, or a bleeding diathesis
17. Therapy for active infection needs to be completed at least 7 days prior to the start of therapy
18. Patients with a known positivity for human immunodeficiency virus (HIV)
19. Patients with active hepatitis B (chronic or acute; HBV) defined as having a positive hepatitis B surface antigen (HbsAg) test at screening. Patients with past or resolved HBV infection (defined as having a negative HbsAg test and a positive antibody to hepatitis B core antigen antibody test) are eligible.
20. Patients with active hepatitis C (HCV) infection defined as having a positive HCV antibody test followed by a positive HCV ribonucleic acid (RNA) test at screening. The HCV RNA test will be performed only for patients who have a positive HCV antibody test. Patients who are positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
21. Serious or non-healing wound, skin ulcer, or non-healing bone fracture
22. Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
23. Albumin <2.8 g/dL or <28 g/L, and without albumin transfusion for ≥7 days prior to screening
24. Unwilling or unable to follow protocol requirements
25. Any live virus vaccine within 30 days prior to the start of therapy
26. Has had an allogenic tissue/solid organ transplant
27. History of another primary malignancy except for:

    1. Malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of investigational product and of relatively low potential risk for recurrence
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    3. Adequately treated carcinoma in situ without evidence of disease
    4. Cancer patients with incidental histologic findings of prostate cancer that, in the opinion of the Investigator, is not deemed to require active therapy (e.g., incidental prostate cancer identified following cystoprostatectomy that is tumor/node/metastasis Stage ≤ pT2N0) may be enrolled, pending discussion and approval by the MM
28. Male or female patients of reproductive potential who are not willing to employ adequate contraception from screening to at least 3 months after the last MP0310 IMP administration
29. Any condition that, in the opinion of the Investigator, would interfere with evaluation of the MP0310 IMP or interpretation of the patient's safety or study results
30. Patient deprived of liberty by a judicial or administrative decision, patient admitted to a social institution or who is under a measure of legal protection, patient hospitalized without consent or who is in an emergency situation
31. Known hypersensitivity or allergy to murine products or any excipients of rituximab (Part C only)
32. Active, severe infections and/or severely immunocompromised state
33. Contraindication against mandatory prophylactic premedication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | From signing of informed consent form (ICF) until 10 weeks following the last dose or start of new anticancer therapy.
  According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Incidence of dose-limiting toxicities (DLTs) | First 21 days of dosing.
  Dose-limiting toxicities will be reviewed as a subset of AEs that occur within the first 21 days of dosing and meet the protocol-specified criteria.
Maximum tolerated dose (MTD) or a tolerated dose below MTD (if MTD is not reached) | From signing of ICF until 10 weeks following the last dose or start of new anticancer therapy.
  Based on occurrence of DLTs within a 3+3 clinical trial design
Recommended expansion dose (RED) | From signing of ICF until 10 weeks following the last dose or start of new anticancer therapy.
  Based on incidence and nature of DLTs, and incidence, nature, and severity of AEs and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Serum concentration - time profiles | 24 months
  Including parameters like maximal serum concentration (Cmax), time at Cmax (Tmax), minimal serum concentration (Cmin)
Area under the serum concentration-time curve (AUC) | 24 months
  Pharmacokinetic (PK) analysis of MP0310
Total clearance (CL) | 24 months
  PK analysis of MP0310
Volume of distribution (Vd), volume at steady state (Vss) | 24 months
  PK analysis of MP0310
Terminal elimination half-life (t1/2) | 24 months
  PK analysis of MP0310
Accumulation ratio | 24 months
  PK analysis of MP0310
Incidence of anti-drug-antibodies | 24 months
  Serum concentration-time profile of anti-drug antibodies
Objective response rate (ORR) | 24 months
  The proportion of participants with confirmed complete response (CR) and partial response (PR) using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and Immunotherapy Response Evaluation Criteria in Solid Tumors (iRECIST)
Disease control rate (DCR) | 24 months
  Stable disease lasting 4 or more weeks following the initiation of MP0310
Duration of response (DoR) | 24 months
  For participants with CR or PR, DOR will be calculated as time from initial response of CR or PR to progressive disease or death.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre Léon Bérard, Lyon
  - Institut Claudius Regaud; Institut Universitaire du Cancer Toulouse Oncopole (IUCT-O), Toulouse
  - Institut Gustave Roussy, Villejuif